CLINICAL TRIAL: NCT02276768
Title: A Phase 1b Clinical Study on the Analgesic Effect of GIC-1001 and GIC-1002 on Visceral Pain Under Rectal Distension and Rectal Sensory Threshold Using the Barostat Method in Male and Female Healthy Volunteers.
Brief Title: Study on Analgesia of GIC-1001 & GIC-1002 on Visceral Pain, Rectal Sensory Threshold Using the Barostat Method
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: gicare Pharma Inc. (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIC1.14.1.02; GCR-P7-403 (Other: Algorithme Pharma Inc.)
Record Dates: First submitted 2014-10-20; First posted 2014-10-28 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Pain; Cancer; Colonic Disease
Keywords: rectal distension; rectal compliance; visceral pain; pain intensity; barostat; distender; VAS (Visual Analog Scale); rectal sensory threshold; analgesia; trimebutine; pain management; peripheral; colon cancer; H2S (hydrogen sulfide)
MeSH Terms: conditions — Pain; Neoplasms; Colonic Diseases; Visceral Pain; Agnosia; Colonic Neoplasms | interventions — trimebutine 3-thiocarbamoylbenzenesulfonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- GIC-1001 mid-dose (Experimental): GIC-1001 , 375 mg TID during 3 consecutive days + a 10th dose in the morning of day 4 (colonoscopy day)
  Interventions: Drug: GIC-1001 375 mg TID
- GIC-1001 high-dose (Experimental): GIC-1001 , 500 mg TID during 3 consecutive days + a 10th dose in the morning of day 4 (colonoscopy day)
  Interventions: Drug: GIC-1001 500 mg TID
- GIC-1002 mid-dose (Active Comparator): GIC-1002 345 mg TID (equimolar to GIC-1001 375 mg) 345 mg TID during 3 consecutive days + a 10th dose in the morning of day 4 (colonoscopy day)
  Interventions: Drug: GIC-1002 345 mg TID (equimolar to GIC-1001 375 mg TID)
- GIC-1002 high-dose (Active Comparator): GIC-1002 460 mg (equimolar to GIC-1001 500 mg) 460 mg TID during 3 consecutive days + a 10th dose in the morning of day 4 (colonoscopy day)
  Interventions: Drug: GIC-1002 460 mg (equimolar to GIC-1001 500 mg)
- Placebo matching GIC-1001 and GIC-1002 (Placebo Comparator): Placebo matching GIC-1001 doses Placebo matching GIC-1002 doses
  Placebo, TID during 3 consecutive days, + a 10 th dose in the morning of day 4 (colonoscopy day)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GIC-1001 375 mg TID — GIC-1001 375 mg TID mid-dose, oral tablet, white-coated, to be taken with water
  Other Names: trimebutine 3-thiocarbamoylbenzenesulfonate , TB-905-02
  Arms: GIC-1001 mid-dose
Drug: GIC-1001 500 mg TID — GIC-1001 500 mg TID high-dose, oral tablet, white-coated, to be taken with water
  Other Names: trimebutine 3-thiocarbamoylbenzenesulfonate , TB-905-02
  Arms: GIC-1001 high-dose
Drug: GIC-1002 345 mg TID (equimolar to GIC-1001 375 mg TID) — GIC-1002 345 mg TID mid-dose, oral tablet, white-coated, to be taken with water
  Other Names: non-H2S releasing tosylate salt
  Arms: GIC-1002 mid-dose
Drug: GIC-1002 460 mg (equimolar to GIC-1001 500 mg) — GIC-1002 460 mg TID high-dose, oral tablet, white-coated, to be taken with water
  Other Names: non-H2S releasing tosylate salt
  Arms: GIC-1002 high-dose
Other: Placebo — Placebo identical and matching active drugs GIC-1001 and GIC-1001
  Other Names: sugar -pill
  Arms: Placebo matching GIC-1001 and GIC-1002

SUMMARY:
This study evaluates colonic analgesia by comparing two novel formulations, GIC-1001 and GIC-1002 with placebo using a barostat distender. The healthy male and female volunteers randomized to one of 5 possible treatments will be exposed to rectal distension following a 3-day treatment TID. The barostat methodology is a well-established and validated way to assess visceral pain. Visceral pain will be evaluated during exposure to varying distender pressures using a visual analog scale.

DETAILED DESCRIPTION:
The objectives of this single center, randomized, double-blinded, placebo-controlled Phase I clinical study include the evaluation of visceral pain intensity under rectal distension following the oral administration of either of two doses of GIC-1001 or of either of two doses of GIC-1002, equimolar to the first formulation, or of placebo in 90 healthy subjects.

The barostat intra-balloon pressure required to elicit pre-defined rectal sensory symptoms (i.e. first sensation, need to defecate, urgency to defecate and pain) will also be determined. Rectal sensory symptom ratings and rectal compliance under increased rectal distension will also be evaluated.

The contribution of hydrogen sulphide (H2S) to the colonic analgesic activity of GIC-1001 by comparison to that of GIC-1002 will be evaluated following steady state pharmacokinetic analysis. To further comprehend the non-linear, U shape dose response curve observed with GIC-1001 in a previous Phase II a trial.

Finally, the safety of GIC-1002 in healthy volunteers will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteer
* A female volunteer must meet one of the following criteria:

Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first dosing, during the study and for at least 30 days after the last dosing or participant is of non-childbearing potential, i.e. surgically sterile or menopausal (at least 1 year without menses)

* Age between 18 to 65 years
* 35.00 kg/m2 ≥ Body Mass Index ≤ 18.50 kg/m2
* Light-, non- or ex-smokers. A light smoker is smoking 2 cigarettes or less per day for at least 3 months before Day 1. An ex-smoker is someone who completely stopped smoking for at least 6 months before Day 1
* Barostat naive or no barostat experience in the year preceding screening
* Clinical laboratory values within the laboratory's stated normal range; or without any clinical significance
* Have no history of clinically significant diseases or evidence of clinically significant findings on physical exam and/or clinical laboratory tests
* Have a normal anorectal area, confirmed by entry digital rectal exam (DRE) and
* Signed dated informed consent form by subject

Exclusion Criteria:

* Pregnant or lactating females
* History of significant hypersensitivity to trimebutine, to sulfur-containing drugs or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose undesired effects
* Diagnosis of Inflammatory Bowel Disease or Irritable Bowel Syndrome
* Criteria for functional bowel disorder (i.e. functional constipation, functional diarrhea and IBS) or abdominal pain, as reported by questionnaire
* Known history of rectosigmoid disease
* Abnormal anorectal findings during entry DRE
* History of abdominal surgery (except appendectomy or cholecystectomy)
* History of gastrointestinal obstruction, any rectal or colon surgery
* Known presence of piles or fissures, peri-anal pathology or any other rectal abnormalities
* Female subjects with history of gynecological surgery (˂ 10 years prior to screening or 1 year for tubal ligation or hysterectomy)
* Known history of, or risk factors for pelvic floor injury
* History of significant gastrointestinal, liver or kidney disease, or surgery
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
* Presence of out-of-range cardiac interval (PR < 110 msec, PR > 220 msec, QRS < 60 msec, QRS >119 msec and QTc > 450 msec for males and > 460 msec for females) on the screening elcetrocardiogram (ECG) or other clinically significant ECG abnormalities
* Use of cysteine, methionine, and other sulfur-containing amino acid supplements in the previous 7 days before day 1 of this study;
* Light-smoker who smokes cigar or is unable to refrain from smoking in the 7 days prior to the housing period and during the housing period of the study
* Known presence of rare hereditary problems of galactose and/or lactose intolerance
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes and strong inducers of CYP enzymes in the previous 28 days before day 1 of this study;
* Regular consumption of any supplement related to bowel movement in the previous 28 days before day 1 of this study
* Positive urine screening of alcohol and/or drugs of abuse
* Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or anti-Hepatitis C Virus (HCV (C)) tests
* Females pregnant according to a positive serum pregnancy test;
* Subjects treated with any Investigational Product in the previous 28 days before Day 1 or who have already participated in this clinical study;
* Prior donation of 50 mL or more of blood in the previous 28 days before Day 1
* Prior total donation of 500 mL or more of blood in the previous 56 days before Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mean visceral pain intensity score following dosing with GIC-1001 375 mg TID | Stage IV, test lasts approximately 20 min.VAS scores collected every 2 minutes at a colorectal distension pressures 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60 mmHg in random order, each maintained for 1 minute.A 1-minute resting period follows between.
  Mean visceral pain intensity score in millimeters (mm) on a 100-mm Visual Analog Scale (VAS) based on 7 measurements collected at increasing rectal distension pressures from 24 to 60 mmHg following the oral administration of the GIC-1001 375 mg TID x 3 days regimen, and comparing it to placebo.

SECONDARY OUTCOMES:
Mean visceral pain intensity score following dosing with GIC-1001 500 mg TID | Stage IV, test lasts approx. 20 min.VAS scores collected every 2 min. at colorectal distension pressures 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60 mmHg in random order, each maintained for 1 minute. A 1-minute resting period follows VAS scoring..
  Mean visceral pain intensity score in mm on a 100-mm VAS based on 7 measurements collected at increasing rectal distension pressures from 24 to 60 mmHg following the oral administration of the GIC-1001 500 mg TID x 3 days regimen, compared to placebo.
Mean visceral pain intensity score following dosing with GIC-1002 345 mg TID and GIC-1002 460 mg TID | Stage IV, test lasts approx. 20 min.VAS scores collected every 2 min. at colorectal distension pressures 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60 mmHg in random order, each maintained for 1 minute. A 1-minute resting period follows VAS scoring.
  Mean visceral pain intensity score in mm on a 100-mm VAS, based on 7 measurements collected at increasing rectal distension pressures from 24 to 60 mmHg following the oral administration of two doses of GIC-1002 (345 mg TID and 460 mg TID x 3 days regimen), compared to placebo.
Barostat pressure required to elicit pre-defined rectal sensory symptoms | Stage III lasts about 15 min.VAS scores collected every 1 minute at increasing colorectal distension pressures: 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56 and 60 mmHg. Each pressure is held for 1 minute for VAS score report. No resting period.
  Barostat intra-balloon pressure in mm Hg required to elicit pre-defined rectal sensory symptoms (i.e. first sensation, need to defecate, urgency to defecate and pain) following the oral administration of GIC-1001 or GIC 1002, respectively at two equimolar doses
Rectal sensory intensity score | Stage III lasts about 15 min.Intensity score recorded every minute at te same time as VAS for rectal sensory compliance...
  Rectal sensory intensity score (i.e. first sensation, need to defecate, urgency to defecate and pain) in mm on a 100-mm VAS following the oral administration of GIC-1001 or GIC-1002, respectively at two equimolar doses.
Rectal compliance under increasing rectal distension | Stage III lasts about 15 min. Overall rectal compliance is calculated over a 15-minute period with pressure increasing sequentially from 4 to 60 mmHg.
  Rectal compliance in ml/mmHg under increased rectal distension following the oral administration of GIC-1001 or GIC-1002, respectively at two equimolar doses.
Contributing hydrogen sulfide analgesia as evaluated by comparing mean visceral pain intensity score differences | Approx. 35 minutes, during total barostat testing period
  Contribution of H2S to GIC-1001 analgesic effects in terms of mean VAS scores differences between GIC-1001 and GIC-1002 at equimolar doses.
Steady state pharmacokinetic AUC (ng/ml/hour) for GIC-1001 and GIC-1002 | Pre-dose, 0, 24, 36, 72, 80 hours post dose
  Steady State pharmacokinetics of GIC-1001 and GIC-1002 at the end of their proposed dosing regimens at pre-dosing times on Treatment Days 1, 2, 3 and on Day 4 of the barostat procedure then 8 hours post-dose .
Number of participants with adverse events | 5 days, from Treatment Day 1 until 24 hours post-barostat distension
  Number of subjects reporting AEs during participation
Number of adverse events | 5 days, from Treatment Day 1 until 24 hours post-barostat distension
  Number of adverse events reported overall
ECG measures | At baseline and post-barostat Day 4
  Safety evaluation: Standard ECG measures
Normality of physical exam | At baseline and post-barostat Day 4
  Safety evaluation: Complete physical examination at both entry and exit
Normality of Proctoscopic examination | On Day 4, prior and post barostat distension
  Safety evaluation: Evaluation of rectum
Standard laboratory measures (biochemistry, hematology, urinalysis) | At screening, pre-dosing (baseline) and post-barostat Day 4
  Safety evaluation: comparative assessment with baseline for all components

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D., Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided